CLINICAL TRIAL: NCT01266421
Title: International Active Surveillance Study of Medication Used for the Treatment of Endometriosis: Visanne Post-approval Observational Study
Brief Title: Visanne Post-approval Observational Study (VIPOS)
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Klaas Heinemann, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2010_03
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Endometriosis
Keywords: DNG; Anemia; Depression
MeSH Terms: conditions — Endometriosis; Anemia; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dienogest (DNG): Women using DNG) for the treatment of endometriosis
- Other approved endometriosis drugs (OAED): Women using hormonal medications approved for endometriosis treatment in all particiapting countries other than DNG.
- Non-approved endometriosis drugs (NAED): Women using hormonal medications not approved for endometriosis treatment in all particiapting countries.

SUMMARY:
The study assesses safety aspects of Dienogest (DNG) 2mg/day (Visanne) used as endometriosis therapy and of other hormonal treatments for endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a common, chronic, gynecological disease characterized by pain and impaired fertility. It causes chronic inflammation, ovarian cyst formation, fibrosis and adhesions. Symptoms seem to respond to decreased circulating estrogen. The mainstay of medical treatment is hormonal induced anovulation and a reduction in endogenous estrogen production.

Medications for endometriosis such as Danazol and GnRH agonists have clinically relevant side-effects limiting treatment duration with these medications to 6-12 months.

Dienogest (DNG) is a 19-nortestosterone derivative progestogen. DNG 2mg/day is a reliable and effective treatment for dysmenorrhea, premenstrual pain, dyspareunia and diffuse pelvic pain associated with endometriosis.

Two important class effects of progestogens are the induction of bleeding disturbances and their influence on mood disturbance. It is not known what influence DNG will have on bleeding disturbances associated with endometriosis, particularly over a longer time frame.

In addition, women who suffer from endometriosis are at high risk of developing depressive symptoms. It is difficult to differentiate if depressive symptoms are causally associated with progestogen use or sequela of the disease process.

This study investigates the safety of DNG for endometriosis with regard to medical interventions for anemia and worsening of depressive symptoms associated with the disease. It is a prospective, controlled, non-interventional cohort study with two cohorts: users of DNG and users of other medications for the treatment of endometriosis. The study will be implemented in several European countries.

ELIGIBILITY:
Inclusion Criteria:

* Women using a newly prescribed regimen for endometriosis (first-time users or switchers or re-starters)
* Women who are willing to participate in this long-term follow-up study

Exclusion Criteria:

* Women who are not cooperative/available for follow-up
* Women with a language barrier

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women using medications for the treatment of endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 27840 (Actual)
Dates: Start 2010-12-07 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-01-26 (Actual)

PRIMARY OUTCOMES:
Anemia | Within 6 years
  Medical intervention for anemia induced by cyclical bleeding disturbances (anemia)
Depression | Within 6 years
  First time occurence of clinically relevant depression, or worsening of existing depression

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, PhD, MD, MBA, Principal Investigator — Center for Epidemiology and Health Research
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Result] Moehner S, Becker K, Lange JA, von Stockum S, Heinemann K. Risk of depression and anemia in users of hormonal endometriosis treatments: Results from the VIPOS study. Eur J Obstet Gynecol Reprod Biol. 2020 Aug;251:212-217. doi: 10.1016/j.ejogrb.2020.05.049. Epub 2020 Jun 2. PMID 32559605
- [Derived] Becker K, Heinemann K, Imthurn B, Marions L, Moehner S, Gerlinger C, Serrani M, Faustmann T. Real world data on symptomology and diagnostic approaches of 27,840 women living with endometriosis. Sci Rep. 2021 Oct 14;11(1):20404. doi: 10.1038/s41598-021-99681-3. PMID 34650132
- [Derived] Heinemann K, Imthurn B, Marions L, Gerlinger C, Becker K, Moehner S, Faustmann T. Safety of Dienogest and Other Hormonal Treatments for Endometriosis in Real-World Clinical Practice (VIPOS): A Large Noninterventional Study. Adv Ther. 2020 May;37(5):2528-2537. doi: 10.1007/s12325-020-01331-z. Epub 2020 Apr 16. PMID 32301063

DOCUMENTS (2):
  • Study Protocol (2011-11-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT01266421/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT01266421/SAP_001.pdf